CLINICAL TRIAL: NCT06625580
Title: Comparison of Ultrasound-Guided Serratus Anterior and Transversus Thoracic Muscle Plane Block Combination Versus Erector Spinae Plane Block for Acute Poststernotomy Pain Management After Cardiac Surgery
Brief Title: Ultrasound-Guided Serratus and Transversus Thoracic Muscle Plane Block Vs. Erector Spinae Plane Block for Acute Poststernotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed E Aydin, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATATURK-Cardiovascular
Record Dates: First submitted 2024-09-22; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-08

CONDITIONS: Pain, Acute; Pain, Chest
MeSH Terms: conditions — Acute Pain; Chest Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ultrasound guided transverse thoracic muscle plane block and serratus anterior plane block (Active Comparator): ultrasound guided transverse thoracic muscle plane block and serratus anterior plane block will be performed with %0.25 bupivacaine
  Interventions: Procedure: transverse thoracic muscle plane and serratus anterior plane block
- ultrasound guided erector spinae plane block (Active Comparator): ultrasound guided erector spinae plane block
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: transverse thoracic muscle plane and serratus anterior plane block — ultrasound guided transverse thoracic muscle plane block and serratus anterior plane block will be performed with 0.25% bupivacaine
  Arms: ultrasound guided transverse thoracic muscle plane block and serratus anterior plane block
Procedure: erector spinae plane block — ultrasound guided erector spinae plane block will be performed with 0.25% bupivacaine
  Arms: ultrasound guided erector spinae plane block

SUMMARY:
Poststernotomy pain represents a complication that can arise following cardiac surgery. Inadequately managed pain has been linked to various adverse outcomes, including myocardial ischemia, cardiac arrhythmias, heightened coagulation tendencies, pulmonary complications, and elevated incidences of delirium and wound infections.

The Erector Spinae Plane (ESP) block, Serratus Anterior Plane (SAP) block, and Transverse Thoracic Muscle Plane (TTMP) block are demonstrated as effective regional anesthesia techniques for sternotomy pain. While these blocks differ in ease of application and efficacy, the optimal analgesic approach for cardiac surgery remains unclear. The aim of this study is to compare the analgesic efficacy of ultrasound-guided SAP and TTMP blocks combination versus ESP block administered alone in patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Surgery with median sternotomy (valvular and coronary surgeries)

Exclusion Criteria:

* Minimal invasive cardiac surgeries
* Revision surgeries (during postoperative 48 hours)
* Redo cardiac surgeries
* Any contraindications for regional anesthesia technique (any allergies for local anesthetics)
* Preoperative chronic opioid usage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Postoperative 48 hours
  postoperative opioid consumption will be recorded for 48 hours

SECONDARY OUTCOMES:
Postoperative Visual Analog Scale | Postoperative 48 hours
  Postoperative Visual Analog Scale assessment will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Enes Aydin, Principal Investigator — Associate Professor
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179
- [Background] Muhammad QUA, Sohail MA, Azam NM, Bashir HH, Islam H, Ijaz R, Aquil S, Mansoor T, Dhakal B, Fatima T, Noor J, Khan AS, Iqbal A, Khatri M, Kumar S. Analgesic efficacy and safety of erector spinae versus serratus anterior plane block in thoracic surgery: a systematic review and meta-analysis of randomized controlled trials. J Anesth Analg Crit Care. 2024 Jan 12;4(1):3. doi: 10.1186/s44158-023-00138-y. PMID 38217050